CLINICAL TRIAL: NCT00711230
Title: A Phase II Randomized, Placebo-Controlled, Multi-Center Study to Evaluate the Safety, Tolerability, Immunogenicity, and Antiretroviral Activity of DermaVir Patch (LC002) in Treatment-Naïve HIV-1-Infected Patients
Brief Title: Repeated DermaVir Immunizations in HIV-1 Infected Treatment-naïve Patients
Acronym: GIEU006
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genetic Immunity (Industry)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DermaVir Phase II; 2007-001955-20 (EudraCT Number)
Record Dates: First submitted 2008-07-04; First posted 2008-07-08 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: HIV Infection
Keywords: HIV; Vaccine; Immune Therapy; DermaVir
MeSH Terms: conditions — HIV Infections | interventions — DermaVir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1: Low dose DermaVir (Experimental): * Dosage: 0.2 mg DNA
  * Dosage form: 1.6 mL DNA/PEIm nanomedicine
  * Administration with 2 DermaPrep patches
  * Frequency: every six weeks
  * Duration: 18 weeks (4 DermaVir treatments)
  Interventions: Biological: DermaVir
- 2: Low dose Placebo (Experimental): * Dosage form: 1.6 mL Placebo
  * Administration with 2 DermaPrep patches
  * Frequency: every six weeks
  * Duration: 18 weeks (4 Placebo treatments)
  Interventions: Biological: Placebo
- 3: Medium dose DermaVir (Experimental): * Dosage: 0.4 mg DNA
  * Dosage form: 3.2 mL DNA/PEIm nanomedicine
  * Administration with 4 DermaPrep patches
  * Frequency: every six weeks
  * Duration: 18 weeks (4 DermaVir treatments)
  Interventions: Biological: DermaVir
- 4: Medium dose Placebo (Experimental): * Dosage form: 1.6 mL Placebo
  * Administration with 4 DermaPrep patches
  * Frequency: every six weeks
  * Duration: 18 weeks (4 Placebo treatments)
  Interventions: Biological: Placebo
- 5: High dose DermaVir (Experimental): * Dosage: 0.8 mg DNA
  * Dosage form: 6.4 mL DNA/PEIm nanomedicine
  * Administration with 8 DermaPrep patches
  * Frequency: every six weeks
  * Duration: 18 weeks (4 DermaVir treatments)
  Interventions: Biological: DermaVir
- 6: High dose Placebo (Experimental): * Dosage form: 6.4 mL Placebo
  * Administration with 8 DermaPrep patches
  * Frequency: every six weeks
  * Duration: 18 weeks (4 Placebo treatments)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: DermaVir
  Other Names: LC002
  Arms: 1: Low dose DermaVir; 3: Medium dose DermaVir; 5: High dose DermaVir
Biological: Placebo — glucose/dextrose
  Arms: 2: Low dose Placebo; 4: Medium dose Placebo; 6: High dose Placebo

SUMMARY:
DermaVir is a synthetic pathogen-like nanomedicine. The active pharmaceutical ingredient is a single plasmid DNA expressing fifteen HIV antigens that assemble to HIV-like particles. These particles are safe; replication, integration and reverse transcription deficient. DermaVir is targeted to Langerhans cells by topical administration with DermaPrep. Langerhans cells with DermaVir migrate to lymph nodes and induce HIV-specific T cells that can kill HIV-infected cells.

GIEU006 is a Phase II randomized, placebo-controlled, dose-finding, double-blinded, multicenter study to assess the safety, tolerability, immunogenicity, and preliminary antiretroviral activity of DermaVir in antiretroviral therapy naïve adults with HIV-infection.

DETAILED DESCRIPTION:
Patients were randomized into one of the following 6 arms:

* Arm 1: Low dose DermaVir (0.2 mg DNA in 2 DermaPrep patches, n=9)
* Arm 2: Low dose Placebo (2 DermaPrep patches, n=3)
* Arm 3: Medium dose DermaVir (0.4 mg DNA in 4 DermaPrep patches, n=9)
* Arm 4: Medium dose Placebo (4 DermaPrep patches, n=3)
* Arm 5: High dose DermaVir (0.8 mg DNA in 8 DermaPrep patches, n=9)
* Arm 6: High dose Placebo (8 DermaPrep patches, n=3) DermaPrep Patch size: 80 cm2. DermaVir Standard Unit per patch is 0.1 mg DNA = 0.8 mL of DermaVir nanomedicine.

The patch sites for immunization are preferably the left or right upper back and left or right upper ventral thigh. The same skin sites should be used for all immunizations.

Immunization schedule (Days): 0, 42, 84, and 126.

The total DermaVir dose:

* Low dose: 0.8 mg DNA
* Medium dose: 1.6 mg DNA
* High Dose: 3.2 mg DNA

DermaVir immunizations were administered over an 18-week period Primary endpoint: 24 weeks Safety follow up: 234 weeks

ELIGIBILITY:
Main inclusion Criteria:

* HIV antibody positive
* Plasma HIV RNA value ≥5,000 copies/mL and ≤ 150,000 c/mL
* Antiretroviral therapy naïve
* Documented CD4+ T-cell count at screening ≥400 cells/mm3

Main exclusion Criteria:

* No skin disease
* No tattoos, or changes in pigmentation at the selected skin immunization sites
* No acute or chronic illness (e.g Hepatitis C)
* No chronic autoimmune diseases
* No treatment with any immune modulating agents

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2008-04; Primary Completion 2011-12 (Actual); Study Completion 2015-01-01 (Actual)

PRIMARY OUTCOMES:
Percent of participants with primary safety endpoint | 24 weeks
  Primary safety endpoint: occurrence of at least two > Grade 3 adverse event including signs/symptoms, lab toxicities, and/or clinical events that is possibly or definitely related to study treatment (as judged by the GIEU006 team, including site clinicians on the team, blinded to treatment arm) any time from the first day of study treatment until 42 days after the last study vaccine administration.

SECONDARY OUTCOMES:
HIV-1 RNA | 24 weeks
CD4+ and CD8+ T-cell counts | 24 weeks
HIV-specific memory T cell responses | 24 weeks
  Measured with Precursors with High Proliferative Capacity (PHPC) assay (Calarota et al. HIV-1-Specific T cell precursors with high proliferative capacity correlate with low viremia and high CD4 counts in untreated individuals. J Immunol 2008;180:5907-15)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Van Lunzen, PhD, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (3):
- Germany (3):
  - ifi-Medizin GmbH at the Asklepios Klinik St. Georg, Hamburg
  - ICH Grindel, Hamburg
  - University Medical Center Hamburg-Eppendorf, Hamburg

REFERENCES:
- [Background] Lisziewicz J, Bakare N, Calarota SA, Banhegyi D, Szlavik J, Ujhelyi E, Toke ER, Molnar L, Lisziewicz Z, Autran B, Lori F. Single DermaVir immunization: dose-dependent expansion of precursor/memory T cells against all HIV antigens in HIV-1 infected individuals. PLoS One. 2012;7(5):e35416. doi: 10.1371/journal.pone.0035416. Epub 2012 May 9. PMID 22590502
- [Background] Lisziewicz J, Toke ER. Nanomedicine applications towards the cure of HIV. Nanomedicine. 2013 Jan;9(1):28-38. doi: 10.1016/j.nano.2012.05.012. Epub 2012 May 30. PMID 22659241
- [Background] Lorincz O, Toke ER, Somogyi E, Horkay F, Chandran PL, Douglas JF, Szebeni J, Lisziewicz J. Structure and biological activity of pathogen-like synthetic nanomedicines. Nanomedicine. 2012 May;8(4):497-506. doi: 10.1016/j.nano.2011.07.013. Epub 2011 Aug 10. PMID 21839051
- [Background] Toke ER, Lorincz O, Somogyi E, Lisziewicz J. Rational development of a stable liquid formulation for nanomedicine products. Int J Pharm. 2010 Jun 15;392(1-2):261-7. doi: 10.1016/j.ijpharm.2010.03.048. Epub 2010 Mar 25. PMID 20347027
- [Background] Lori F. DermaVir: a plasmid DNA-based nanomedicine therapeutic vaccine for the treatment of HIV/AIDS. Expert Rev Vaccines. 2011 Oct;10(10):1371-84. doi: 10.1586/erv.11.118. PMID 21988301
- [Background] Somogyi E, Xu J, Gudics A, Toth J, Kovacs AL, Lori F, Lisziewicz J. A plasmid DNA immunogen expressing fifteen protein antigens and complex virus-like particles (VLP+) mimicking naturally occurring HIV. Vaccine. 2011 Jan 17;29(4):744-53. doi: 10.1016/j.vaccine.2010.11.019. Epub 2010 Nov 23. PMID 21109034
- [Background] Calarota SA, Weiner DB, Lori F, Lisziewicz J. Induction of HIV-specific memory T-cell responses by topical DermaVir vaccine. Vaccine. 2007 Apr 20;25(16):3070-4. doi: 10.1016/j.vaccine.2007.01.024. Epub 2007 Jan 22. PMID 17292518
- [Background] Lisziewicz J, Trocio J, Whitman L, Varga G, Xu J, Bakare N, Erbacher P, Fox C, Woodward R, Markham P, Arya S, Behr JP, Lori F. DermaVir: a novel topical vaccine for HIV/AIDS. J Invest Dermatol. 2005 Jan;124(1):160-9. doi: 10.1111/j.0022-202X.2004.23535.x. PMID 15654970
- [Background] Lori F, Trocio J, Bakare N, Kelly LM, Lisziewicz J. DermaVir, a novel HIV immunisation technology. Vaccine. 2005 Mar 18;23(17-18):2030-4. doi: 10.1016/j.vaccine.2005.01.004. PMID 15755566
- [Background] Lisziewicz J, Trocio J, Xu J, Whitman L, Ryder A, Bakare N, Lewis MG, Wagner W, Pistorio A, Arya S, Lori F. Control of viral rebound through therapeutic immunization with DermaVir. AIDS. 2005 Jan 3;19(1):35-43. doi: 10.1097/00002030-200501030-00004. PMID 15627031
- See also: Genetic Immunity's homepage — http://www.geneticimmunity.com
- See also: DermaVir for initial treatment of HIV-infected subjects demonstrates preliminary safety, immunogenicity and HIV-RNA reduction versus placebo immunization — http://hivandhepatitis.com/2010_conference/AIDS2010/docs/post/lunzen.pdf